CLINICAL TRIAL: NCT06825416
Title: Multicenter, Randomized, Double-blind, Active-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of SHR-2004 Injection in the Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Knee Arthroplasty
Brief Title: Phase III Clinical Study of SHR-2004 Injection in Preventing Venous Thromboembolism in Patients Undergoing Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SHR-2004-301
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Prevention of Arterial and Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — enoxaparin sodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Drug: SHR-2004 injection; Drug: Enoxaparin sodium injection placebo; Drug: SHR-2004 placebo
- Group B (Experimental)
  Interventions: Drug: SHR-2004 injection; Drug: Enoxaparin sodium injection placebo; Drug: SHR-2004 placebo
- Group C (Active Comparator)
  Interventions: Drug: Enoxaparin sodium injection; Drug: SHR-2004 placebo

INTERVENTIONS:
Drug: SHR-2004 injection — SHR-2004 injection in low dose.
  Arms: Group A
Drug: SHR-2004 injection — SHR-2004 injection in high dose.
  Arms: Group B
Drug: Enoxaparin sodium injection — Enoxaparin sodium injection.
  Arms: Group C
Drug: Enoxaparin sodium injection placebo — Enoxaparin sodium injection placebo.
  Arms: Group A; Group B
Drug: SHR-2004 placebo — SHR-2004 placebo in low dose.
  Arms: Group B; Group C
Drug: SHR-2004 placebo — SHR-2004 placebo in high dose.
  Arms: Group A; Group C

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of SHR-2004 in preventing venous thromboembolism after elective unilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the research procedures and methods, volunteer to participate in this trial, and sign the informed consent form in writing;
2. Planned elective schedule total knee arthroplasty (TKA) patients;
3. Men or women who are ≥ 18 years old and < 80 years old on the day of signing the informed consent form.

Exclusion Criteria:

1. Unable to receive CT angiography of both lower limbs;
2. Malignant tumor within one year of the screening;
3. Myocardial infarction, transient ischemic attack or ischemic stroke occurred within 6 months of the screening;
4. Any medical history that may increase the risk of bleeding or any conditions that the investigator considers to increase the risk of bleeding;
5. History of drug abuse;
6. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1167 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of asymptomatic deep vein thrombosis (DVT) | Day 12.
Incidence of non-fatal pulmonary embolism (PE) | Day 12.

SECONDARY OUTCOMES:
Adverse events (AEs) | Day 65.
Bleeding events | Day 12.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fourth Medical Center of Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Xiangya Hospital, Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided